CLINICAL TRIAL: NCT04619043
Title: Evaluation of a Prescription Model to Customize Passive-Dynamic Ankle-Foot Orthoses for Persons Post-Stroke
Brief Title: Understanding the Effects of Quantitatively-Prescribing Passive-Dynamic Ankle-Foot Orthosis Bending Stiffness for Individuals Post-Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 395018-16
Record Dates: First submitted 2020-10-23; First posted 2020-11-06 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Gait, Hemiplegic
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Ankle Orthotic (Experimental): The participant will wear two different ankle orthotics, their currently prescribed orthotic and the experimental orthotic.
  Interventions: Device: Ankle Orthotic

INTERVENTIONS:
Device: Ankle Orthotic

SUMMARY:
When people walk, their ankle joints help to hold them upright and move them forward. Ankle braces are often given to people who have had a stroke to help their ankle joints work properly. The investigators have developed a method to design and make a special type of ankle brace that allows the investigators to control every characteristic of the ankle brace, allowing the investigators to customize the ankle brace to fit and function just the way the investigators want it to. The investigators think that ankle braces customized to meet the needs of each individual person will help the participants walk better. The investigators have also developed a prescription model that tells the investigators how to customize these ankle braces to address different levels of two common impairments experienced by people post stroke -decreased ability to move the ankle joint and weakened calf muscles. The purpose of this study is to test the prescription model to see if wearing the ankle brace customized based on the prescription model improves people's ability to walk. To accomplish this goal, the investigators will first measure each person's ability to move his/her ankle joint and the strength of his/her calf muscles. The investigators will put this information in to the prescription model to determine how to customize the ankle brace for each person. The investigators will then use the method developed to make the customized ankle brace. Finally, the investigators will measure how each person walks in the ankle brace customized just for the participants. This study will allow the investigators to validate and/or refine the prescription model and teach the investigators how persons post-stroke adapt to walking in ankle braces with different characteristics.

ELIGIBILITY:
Inclusion Criteria:

* 21-85 years of age
* chronic hemiparesis stroke (> 6 months post stroke)
* prescribed an AFO by a clinician
* able to walk for at least two minutes without assistance from another person
* adequate paretic dorsiflexion range-of-motion (RoM ≥ 12°)
* plantar flexor strength deficits (peak paretic plantar flexion moment in gait at least 0.15 Nm/kg lower than the mean speed-matched, height normalized value from our normative database)

Exclusion Criteria:

* cerebellar signs (ataxic ("drunken") gait or decreased coordination during rapid alternating hand or foot movements)
* neurologic conditions other than stroke
* more than one stroke
* sensorimotor neglect
* intermittent claudication
* inability to walk outside the home prior to the stroke
* total joint replacement and orthopedic problems in the lower limbs or spine that limit walking
* coronary artery bypass graft or myocardial infarction within past 3 months
* unexplained dizziness in last 6 months
* cannot understand spoken instruction, communicate with the investigators
* walk for 2 minutes at a self-selected speed without assistance from another person (assistive device allowed)
* must have a resting heart rate between 40-100 beats per minute and a resting blood pressure between 90/60 to 170/90.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Peak Plantar Flexion Moment | 4 weeks
  The peak plantar flexion moment (Newton - meters per degree) will be measured at 0, 2, and 4 weeks via an instrumented gait analysis while the participant walks at their self-selected walking speed wearing their ankle brace.
Step Length | 4 weeks
  Step Length (meters) will be measured via an instrumented gait analysis 0, 2, and 4 weeks while the participant walks at their self-selected walking speed wearing their ankle brace.
Step Ratio | 4 weeks
  Step ratio (unitless) will be measured via an instrumented gait analysis 0, 2, and 4 weeks while the participant walks at their self-selected walking speed wearing their ankle brace.
Propulsion Impulse Ratio | 4 weeks
  Propulsion Impulse Ratio (unitless) will be measured via an instrumented gait analysis 0, 2, and 4 weeks while the participant walks at their self-selected walking speed wearing their ankle brace.
Ankle Power | 4 weeks
  Ankle Power (Work) will be measured via an instrumented gait analysis 0, 2, and 4 weeks while the participant walks at their self-selected walking speed wearing their ankle brace.
Propulsion Force | 4 weeks
  Propulsion Force (Newtons) will be measured via an instrumented gait analysis 0, 2, and 4 weeks while the participant walks at their self-selected walking speed wearing their ankle brace.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware STAR Campus, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olney SJ, Griffin MP, McBride ID. Temporal, kinematic, and kinetic variables related to gait speed in subjects with hemiplegia: a regression approach. Phys Ther. 1994 Sep;74(9):872-85. doi: 10.1093/ptj/74.9.872. PMID 8066114
- [Background] Nadeau S, Gravel D, Arsenault AB, Bourbonnais D. Plantarflexor weakness as a limiting factor of gait speed in stroke subjects and the compensating role of hip flexors. Clin Biomech (Bristol). 1999 Feb;14(2):125-35. doi: 10.1016/s0268-0033(98)00062-x. PMID 10619100
- [Background] Olney SJ, Richards C. Hemiparetic gait following stroke. Part i: Characteristics. Gait Posture 4:136-148, 1996
- [Background] Peterson CL, Kautz SA, Neptune RR. Muscle work is increased in pre-swing during hemiparetic walking. Clin Biomech (Bristol). 2011 Oct;26(8):859-66. doi: 10.1016/j.clinbiomech.2011.04.010. Epub 2011 May 24. PMID 21605927
- [Background] Peterson CL, Hall AL, Kautz SA, Neptune RR. Pre-swing deficits in forward propulsion, swing initiation and power generation by individual muscles during hemiparetic walking. J Biomech. 2010 Aug 26;43(12):2348-55. doi: 10.1016/j.jbiomech.2010.04.027. Epub 2010 May 13. PMID 20466377
- [Background] Mulroy S, Gronley J, Weiss W, Newsam C, Perry J. Use of cluster analysis for gait pattern classification of patients in the early and late recovery phases following stroke. Gait Posture. 2003 Aug;18(1):114-25. doi: 10.1016/s0966-6362(02)00165-0. PMID 12855307
- [Background] Knarr BA, Higginson JS, Binder-Macleod SA. Validation of an adjustment equation for the burst superimposition technique in subjects post-stroke. Muscle Nerve. 2012 Aug;46(2):267-9. doi: 10.1002/mus.23431. PMID 22806377
- [Derived] Skigen JT, Koller CA, Nigro L, Reisman DS, McKee Z, Pinhey SR, Henderson A, Wilken JM, Arch ES. Customized passive-dynamic ankle-foot orthoses can improve walking economy and speed for many individuals post-stroke. J Neuroeng Rehabil. 2024 Jul 29;21(1):126. doi: 10.1186/s12984-024-01425-7. PMID 39069629
- [Derived] Koller C, Reisman D, Richards J, Arch E. Understanding the effects of quantitatively prescribing passive-dynamic ankle-foot orthosis bending stiffness for individuals after stroke. Prosthet Orthot Int. 2021 Aug 1;45(4):313-321. doi: 10.1097/PXR.0000000000000012. PMID 33840749